CLINICAL TRIAL: NCT04772274
Title: A Randomised, Double-blind, Three-arm, Parallel Group, Single-dose Study to Compare the Pharmacokinetics, Safety, Tolerability, and Immunogenicity of Ustekinumab (SB17, EU Sourced Stelara®, and US Sourced Stelara®) in Healthy Subjects
Brief Title: A Study to Compare SB17 (Proposed Ustekinumab Biosimilar) to European Union (EU) Sourced Stelara and United States of America (US) Sourced Stelara in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SB17-1001
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Healthy
MeSH Terms: interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SB17 (Experimental): SB17 (proposed ustekinumab biosimilar)
  Interventions: Drug: Ustekinumab
- EU Stelara (Active Comparator): EU sourced Stelara (ustekinumab)
  Interventions: Drug: Ustekinumab
- US Stelara (Active Comparator): US sourced Stelara (ustekinumab)
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — 45 mg, single-dose

SUMMARY:
This is a randomised, double-blind, three-arm, parallel group, single-dose study to evaluate the pharmacokinetics, safety, tolerability, and immunogenicity of SB17 compared to EU sourced Stelara® and US sourced Stelara® in healthy subjects

DETAILED DESCRIPTION:
This study is a randomised, double-blind, three-arm, parallel group, single-dose study. A total of 201 healthy subjects aged 18-55 years will be randomised 1:1:1 to receive a single dose of either SB17, EU sourced Stelara®, or US sourced Stelara®. All investigational products (IPs) will be administered subcutaneously in the abdomen.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, aged 18-55 years (inclusive) on the day of signing the informed consent.
2. Have a body weight between 60.0-90.0 kg (inclusive) and a body mass index (BMI) between 19.0-29.9 kg/m2 (inclusive) at Screening and Day -1.
3. Have 12-lead electrocardiogram (ECG) results without clinically significant abnormal findings confirmed by the Investigator at Screening and Day -1.
4. Have vital sign results without clinically significant abnormal findings confirmed by the Investigator at Screening and Day -1.
5. Have physical examination results without clinically significant abnormal findings confirmed by the Investigator at Screening and Day -1.
6. Female subjects who are not pregnant or nursing at Screening and Day -1, and subjects who are not planning to become pregnant during study period and until 15 weeks after the IP administration.
7. Female subjects of non-childbearing potential, defined as one of the following:

   1. At least 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., appropriate age) and follicle-stimulating hormone (FSH) in the range for menopausal female confirmed by blood test according to current local standards at Screening
   2. Those with history of hysterectomy or surgical removal of both ovaries. Documentation of surgical procedure performed at least 90 days prior to Screening or documentation of physical examination is required for confirmation of surgical sterilisation OR Female subjects of childbearing potential or male subjects with their (respectively male or childbearing female) partners who agree to use at least two forms of appropriate contraception method (e.g., established use of oral, injected, intravaginal, transdermal, or implanted hormonal contraceptive, placement of an intrauterine device or intrauterine hormone-releasing system, physical barrier [Note: Female condom and male condom should not be used together]) from Screening until 15 weeks after the IP administration. Vasectomy alone will be allowed for male subjects and female subjects of childbearing potential with a sole vasectomised male partner. Vasectomised subjects or partners should be medically confirmed for sterilisation. True abstinence alone will be allowed if this is in line with the preferred and usual lifestyle of the subject, or for subjects who do not have a partner. Contraceptive methods do not apply for subjects whose partner is on the same gender.
8. Willing and able to comply with the scheduled visits, treatment plan, clinical laboratory tests, and other study procedures including lifestyle considerations.
9. Provision of signed and dated written informed consent, which must be obtained prior to any study-related procedures being performed.
10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted.

Exclusion Criteria:

1. Have a history and/or current presence of clinically significant atopic allergy, hypersensitivity, or allergic reactions (either spontaneous or following drug administration), also including known or suspected clinically relevant drug hypersensitivity to ustekinumab or to any of the excipients.
2. Have a history of and/or current clinically significant gastrointestinal, renal, hepatic, cardiovascular, haematological, neurologic (including reversible posterior leukoencephalopathy syndrome), metabolic (including known diabetes mellitus), psychiatric disorder, drug or alcohol abuse, or allergic disease excluding mild asymptomatic seasonal allergies.
3. Have a history of significant respiratory disorder (including asthma, non-infectious pneumonia).
4. Have a history of malignancy (including lymphoma, leukaemia, and skin cancer).
5. Have either active or latent tuberculosis (TB) as indicated by a positive test result for Mycobacterium tuberculosis at Screening or who have a history of TB.
6. Have a history of serious infection (associated with hospitalisation and/or which required IV antibiotics) within 180 days prior to Randomisation.
7. Have a history of invasive systemic fungal infections (e.g., histoplasmosis) or other opportunistic infections judged relevant by the Investigator.
8. Have a clinically significant active infection (bacterial, viral, or fungal) within 28 days prior to Randomisation.
9. Have any systemic or local infection, a known risk for developing sepsis and/or a known active inflammatory process at Screening or Day -1.
10. Have previously been exposed to ustekinumab (Stelara® and its biosimilar).
11. Have previously been exposed to a monoclonal antibody or fusion protein within 270 days (other than ustekinumab) prior to Randomisation and/or there is confirmed evidence or clinical suspicion of immunogenicity from previous exposure to a monoclonal antibody or fusion protein.
12. Have previously been exposed to an immunosuppressive agent or biological agent (any other than a monoclonal antibody or fusion protein) within 120 days prior to Randomisation.
13. Have received Bacillus of Calmette and Guerin (BCG) vaccine within 12 months prior to Randomisation or will require BCG vaccine within 12 months after the IP administration.
14. Have received live vaccine(s) (other than the BCG vaccine) within 30 days prior to Randomisation or will require live vaccine(s) within 15 weeks after the IP administration.
15. Have a personal or family history of prolonged QT interval syndrome or Torsade de Pointes, or family history of sudden death.
16. Have any of the following abnormal laboratory test results at Screening or Day -1.

    1. Serum C-reactive protein ≥ 1.5 × upper limit of normal (ULN)
    2. Serum alanine transaminase (ALT) and/or aspartate transaminase (AST) ≥ 1.5 × upper limit of normal (ULN).
    3. Any other laboratory abnormalities assessed as clinically significant by the Investigator
17. Have a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antibody at Screening.
18. Have a history of immunodeficiency.
19. Have had surgery (including invasive dental treatment or dental surgery) within 90 days prior to Randomisation, and/or plan to have an operation during the study period.
20. Have had a history and/or current presence of an illness within 14 days prior to Randomisation that is classified as clinically significant by the Investigator.
21. Have a history of and/or current Coronavirus Disease-2019 (COVID-19) defined as one of the following:

    1. Positive test result for COVID-19 by an antigen test for SARS-CoV-2 at Day -1. (An antigen test for Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) will be performed twice at Day -1. Pharyngeal swab specimen will be collected separately for each test. If any of two tests are positive, the subject will be excluded from the study.)
    2. Signs and symptoms consistent with COVID-19 (e.g., fever, dry cough, dyspnea, sore throat, or fatigue) 30 days prior to Randomisation.
    3. Have had a positive test result for COVID-19 confirmed by SARS-CoV-2 detection using real-time reverse transcriptase polymerase chain reaction (RT-PCR).
    4. Had a severe course of COVID-19 (e.g., extracorporeal membrane oxygenation (ECMO) or mechanically ventilate).
22. Have smoked more than 10 cigarettes, 2 cigars, or 2 pipes per day within 90 days prior to Randomisation.
23. Have regular consumption of alcoholic beverages that exceeds 14 units per week (1 unit = 12 g of pure alcohol).
24. Have a positive urinary drug screening result or alcohol breath test result at Screening or Day -1.
25. Have taken any prescription medicine or over-the-counter medicines (except paracetamol) within 30 days prior to Randomisation that might have an effect on the objectives of the study in the opinion of the Investigator.
26. Have donated > 100 mL blood or plasma within 28 days prior to Randomisation.
27. Have participated in another study with an investigational drug within 60 days prior to Randomisation or are currently participating in or intending to participate in another clinical study of an investigational drug before completion of all scheduled evaluations in this clinical study.
28. Subjects who, in the opinion of the Investigator, are not likely to complete the study for whatever reason.
29. Subject who is the Investigator or any sub-Investigator, research assistant, pharmacist, study coordinator, other staff, or relative thereof directly involved in the conduct of the clinical study.
30. Vulnerable subjects (e.g., persons kept in detention).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
AUCinf | Day 1 to Day 99
  Area under the concentration-time curve from time zero to infinity
Cmax | Day 1 to Day 99
  Maximum serum concentration

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Day 1 to Day 99
  Experience at least 1 TEAE
Incidence of serious adverse events (SAEs) | Day 1 to Day 99
  Experience at least 1 SAE
Incidence of anti-drug antibodies (ADAs) | Day 1 to Day 99
  Incidence of ADAs to ustekinumab

CONTACTS AND LOCATIONS:
Overall Officials: Hakim Charfi, MD, Principal Investigator — Biotrial Rennes
Locations (1):
- Biotrial Rennes, Rennes, France